CLINICAL TRIAL: NCT07366632
Title: A Phase I, International, Multicenter Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Dose of BL0175 Injection Compared With a Single Dose of Fulvestrant Injection in Postmenopausal Women
Brief Title: A Study of Single Dose of BL0175 in Postmenopausal Women
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Best-Link Bioscience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BL0175-101
Record Dates: First submitted 2026-01-13; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Postmenopausal Women
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BL0175 250mg (Experimental)
  Interventions: Drug: BL0175
- Fulcestrant 250mg (Active Comparator)
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: BL0175 — BL0175 is a polymer-drug conjugate, composed of a steroidal estrogen receptor antagonist fulvestrant covalently linked to a PEG-modified poly- polymer via a peptide based cleavable linker
  Arms: BL0175 250mg
Drug: Fulvestrant — Fulvestrant Injection has been marked in many country and regions for the treatment of women who have been through menopause with:
  * hormone receptor (HR) positive, human epidermal growth factor receptor 2 (HER2) negative, locally advanced or metastatic breast cancer who have not been previously treated with endocrine therapy.
  * HR positive, locally advanced or metastatic breast cancer who have progressive disease following prior endocrine (anti-oestrogen or aromatase inhibitor) therapy.
  Fulvestrant stops some of the actions of oestrogen within the body. Oestrogen is a female sex hormone that may help cancer cells grow in women with breast cancer.
  Arms: Fulcestrant 250mg

SUMMARY:
The goal of this clinical trial is to learn the safety and PK of the single dose of BL0175 Injection in postmenopausal women and to compare that with a single dose of Fulvestrant Injection. The main questions it aims to answer are:

* What medical problems do participants have when using drug BL0175?
* How long can BL0175 remain in your blood? Participants will receive a single dose of drug BL0175 or a single dose of Fulvestrant Injection in a randomized method

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study, be able to understand the requirements of a clinical study, and sign informed consent form.
2. Postmenopausal female participants aged ≥ 18 years old.
3. Body weight ≥ 45kg and body mass index (BMI= weight/height2) scores ≥ 18 kg/m2 and ≤ 35 kg/m2.
4. Participants with laboratory tests, physical examinations, vital signs, and electrocardiogram (ECG) results judged by the investigator as normal or abnormal with no clinical significance (NCS).

Exclusion Criteria:

1. Participants with a history or current presence of any cardiovascular, gastrointestinal, endocrine, hematological, hepatic, immunological, metabolic, urinary, pulmonary, neurological, dermatological, psychiatric, renal, and/or other major diseases that are considered clinically significant by the investigator.
2. A history of allergy to fulvestrant, alcohol, castor oil, benzyl alcohol, benzyl benzoate or any other comparable or similar products, or prone to allergic reactions (such as: prone to angioedema, urticaria, asthma, rash, etc.), or history of allergy to two or more drugs (or foods).
3. Participants with current concomitant sciatica, neuralgia, or peripheral neuropathy.
4. History of allogeneic transplantation of organs, bone marrow or stem cell.
5. Active infection, a known history of hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection or screening for infectious disease (HBsAg, hepatitis C virus antibody [HCV-Ab], or human immunodeficiency virus antigen/antibody [HIV-Ag/Ab]) during the screening period is positive.
6. Unable to refrain from or anticipate the use of any prescription medications not for the treatment of concomitant diseases within 4 weeks prior to administration, or any over-the-counter drugs (including but not limited to Chinese herbal medicines, compound preparations of Chinese herbal medicines, health products, etc.) not for the treatment of concomitant diseases within 2 weeks prior to administration.
7. Participants who are vaccinated within 14 days prior to dosing administration.
8. Those who donated plasma or blood within 12 weeks prior to the dosing administration or donated or lost blood 400 mL or more within 12 weeks prior to the dosing administration, or plan to donate during the study.
9. Any history of coagulation dysfunction, bleeding diathesis (e.g., disseminated intravascular coagulation, coagulation factor deficiencies), long-term anticoagulant therapy (excluding antiplatelet therapy and low-dose warfarin), active bleeding (such as gastrointestinal bleeding), or clinically significant thrombocytopenia.
10. Intolerance to / fear of venipuncture, needles, or blood collection difficulties (such as poor vascular conditions, fear of blood collection, needle dizziness, etc.).
11. Those who underwent major surgery within 4 weeks before screening, or plan to undergo major surgery during the study.
12. Those who have taken/used investigational drugs, vaccines or devices within the 4 weeks or 5 half-lives of investigational drug (whichever is longer) prior to the dosing administration.
13. Participants who with a history of alcoholism, or with a history of alcohol abuse within 3 months prior to screening (by self-declaration) > 14 alcohol units per week (1 alcohol unit is about equal to 50° white wine 35 mL or 5° beer 350 mL or wine 150 mL). Participants are unable/unwilling to refrain from alcohol, or strenuous exercise 48 hours prior to each study visit.
14. Participants who with a history of drug abuse or drug dependence, or those who have used illicit drugs within 1 year prior to screening.
15. Positive alcohol or drug screen results at Baseline.
16. Those who are determined by the investigator to be ineligible for other reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v6.0 | from Day 1 to Day 57

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameters-Maximum concentration (Cmax) of fulvestrant | From Day 1 to Day 197
Serious adverse events (SAE) that related to investigational product | up to 197 days
Pharmacokinetics (PK) parameters-Area under the concentration curve (AUC) of fulvestrant | From Day 1 to Day 197
Half-life (t1/2)of fulvestrant | From Day 1 to Day 197